CLINICAL TRIAL: NCT00328601
Title: Assessment of Efficacy and Safety of Thioctic Acid in the Oral Treatment of Symptomatic Diabetic Neuropathy (SYDNEY 2) Randomised, Double-blind,Placebo-controlled Multicentre Trial With 4 Parallel Groups
Brief Title: Assessment of Efficacy and Safety of Thioctic Acid in the Oral Treatment of Symptomatic Diabetic Neuropathy (SYDNEY 2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D-20557-3258
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2008-07

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Thioctic Acid

INTERVENTIONS:
Drug: Thioctic Acid

SUMMARY:
The primary objective of the trial is to determine the optimal dose of orally (tablet) administered thioctic acid in the treatment of symptoms of diabetic polyneuropathy (dPNP). It is expected that at least one of the three dosages to be tested (600, 1200, or 1800 mg tablets) of orally administered thioctic acid improves the symptoms of dPNP as compared to placebo.

Secondary objectives are evaluations of other variables pertinent to dPNP, safety, and tolerability.

DETAILED DESCRIPTION:
Following a screening visit, patients will receive placebo oral for 7 days. Eligible patients with chronic symptoms will then randomly be assigned to one of 4 treatment groups and treated with trial medication for 5 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus (Type I or II), as defined by the American Diabetes Association, 1997, lasting 1 year.
2. Patient must have a symmetric sensory-motor peripheral polyneuropathy of at least stage 2 attributable to diabetes mellitus following a thorough evaluation for other causes of neuropathy.
3. HbA1C < 10%.
4. TSS > 7.5 points.
5. NISLL > 2 points.
6. Pain sensation (according to pin-prick sensitivity test) absent or decreased (NIS item 35 1).
7. Age range: 18 to 74 years. Inclusion criteria prior to randomisation
8. The TSS must be > 5 points
9. The TSS range (maximum TSS minus minimum TSS during the run-in phase) must be less than 3 points to avoid inclusion of patients with rapidly oscillating symptoms.
10. At least 1 of the 4 symptoms of the TSS must have occurred continuously over the last 3 months.
11. Lack of compliance, i.e. below 85% or above 115% (Accordingly, 6 daily doses taken of the 7 daily doses scheduled for Phase A would be acceptable).

Exclusion Criteria:

Lack of suitability for the trial:

1. Proximal asymmetric neuropathy, cranial neuropathies, truncal radiculopathy, diabetic plexopathies, or acute or active mononeuropathies (including cranial neuropathies, post-herpes neuralgias, etc.), with the exception of carpal tunnel syndrome (CTS) or tardy ulnar neuropathy (TUN) or both.
2. Neuropathy of any cause other than diabetes mellitus which might interfere with the assessment of the severity of dPNP.
3. Other neurologic diseases that may produce weakness, sensory loss, or autonomic symptoms or test abnormality.
4. Myopathy of any cause.
5. Peripheral vascular disease severe enough to cause intermittent claudication or ischemic ulcers or limb ischemia.
6. Patients with proliferating retinopathy requiring immediately therapy and impending blindness.
7. Psychiatric, psychological, or behavioural symptoms that would interfere with the patient's ability to participate in the trial.
8. Patients with any active neoplastic disease except basal cell carcinoma.
9. Patients with atrial fibrillation unless controlled and stabilised by medication.
10. Patients with clinically significant cardiac, pulmonary, gastrointestinal, haematological, or endocrine disease (other than diabetes) that may confound interpretation of the study results or prevent the patient from completing the study.
11. Patients who have had organ transplants of any kind.
12. Patients with significant hepatic or renal disease (ASAT, ALAT or GGT >2 times normal, serum creatinine >1.8 mg/dL (>159 mmol/l) for males or >1.6 mg/dL (>141 mmol/l) for females).
13. Patients with a recent history (within last 12 months) of drug or alcohol abuse.
14. Use of any investigational drug (participation in a clinical trial) within last 1 month.
15. History of severe or anaphylactic reaction to drugs, sulfur or biologic products.
16. Recent (within last 3 months) ketoacidosis or hypoglycaemia, necessitating hospital admission.
17. Antioxidant therapy (vitamins E > 400 IU, C > 200 mg, and beta-Carotene > 30 mg) or pentoxyphylline within last 1 month before start of trial.
18. Use of thioctic acid (> 50 mg), evening primrose oil or any other gamma-linolenic acid containing substance within the last 3 months.
19. Continued use of medications listed in section 6.2.3.
20. Bilateral sural nerve biopsies.
21. Existing foot ulcers.

    Safety concerns:
22. Pregnant or lactating females: Pregnancy as evidenced by positive b-hCG-test at screening visit or by testing performed at the study site on demand, or women of child-bearing potential not using adequate contraception.
23. History of allergic reaction to the study medication or its excipients.

    Administrative reasons:
24. Informed Consent is not signed or the patient has not complete competence to co-operate.
25. Any language barriers that can affect adequate understanding.
26. Anticipated non-availability for study visits/procedures.
27. Vulnerable subjects (such as persons kept in detention)

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170
Dates: Start 2005-02; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Dan Ziegler, Prof., Principal Investigator — German Diabetes Research Institute, Heinrich Heine University, Auf'm Hennekamp 65, D-40225 Düsseldorf, Germany
Locations (5):
- Israel (2):
  - Wolfson Medical Center, Diabetes Unit, Holon
  - Haddassah Medical Center Ein Kerem, Diabetes Unit, Jerusalem
- Russia (3):
  - Chair of Nervous Diseases of IM Sechenov Moscow Medical Academy at City Clinical Hospital, Moscow
  - Chair of Endocrinology and Diabetology of Russian Medical Academy of Postgraduate Education at Central Clinical Hospital of Ministry of Communication RF, Moscow
  - Federal Centre of Medical Social Expertise and Rehabilitation of Invalids, Centre Diabetic Food, Moscow

REFERENCES:
- [Background] Wang PH, Lau J, Chalmers TC. Meta-analysis of effects of intensive blood-glucose control on late complications of type I diabetes. Lancet. 1993 May 22;341(8856):1306-9. doi: 10.1016/0140-6736(93)90816-y. PMID 8098449
- [Background] Inzucchi SE. Oral antihyperglycemic therapy for type 2 diabetes: scientific review. JAMA. 2002 Jan 16;287(3):360-72. doi: 10.1001/jama.287.3.360. PMID 11790216
- [Background] Collins SL, Moore RA, McQuayHJ, Wiffen P. Antidepressants and anticonvulsants for diabetic neuropathy and postherpetic neuralgia: a quantitative systematic review. J Pain Symptom Manage. 2000 Dec;20(6):449-58. doi: 10.1016/s0885-3924(00)00218-9. PMID 11131263
- [Background] Jarvis B, Coukell AJ. Mexiletine. A review of its therapeutic use in painful diabetic neuropathy. Drugs. 1998 Oct;56(4):691-707. doi: 10.2165/00003495-199856040-00016. PMID 9806111
- [Background] Rains C, Bryson HM. Topical capsaicin. A review of its pharmacological properties and therapeutic potential in post-herpetic neuralgia, diabetic neuropathy and osteoarthritis. Drugs Aging. 1995 Oct;7(4):317-28. doi: 10.2165/00002512-199507040-00007. PMID 8535059
- [Background] Cameron NE, Cotter MA. The relationship of vascular changes to metabolic factors in diabetes mellitus and their role in the development of peripheral nerve complications. Diabetes Metab Rev. 1994 Oct;10(3):189-224. doi: 10.1002/dmr.5610100302. No abstract available. PMID 7835170
- [Background] Smith AR, Shenvi SV, Widlansky M, Suh JH, Hagen TM. Lipoic acid as a potential therapy for chronic diseases associated with oxidative stress. Curr Med Chem. 2004 May;11(9):1135-46. doi: 10.2174/0929867043365387. PMID 15134511
- [Background] Cameron NE, Cotter MA, Archibald V, Dines KC, Maxfield EK. Anti-oxidant and pro-oxidant effects on nerve conduction velocity, endoneurial blood flow and oxygen tension in non-diabetic and streptozotocin-diabetic rats. Diabetologia. 1994 May;37(5):449-59. doi: 10.1007/s001250050131. PMID 8056181
- [Background] Nagamatsu M, Nickander KK, Schmelzer JD, Raya A, Wittrock DA, Tritschler H, Low PA. Lipoic acid improves nerve blood flow, reduces oxidative stress, and improves distal nerve conduction in experimental diabetic neuropathy. Diabetes Care. 1995 Aug;18(8):1160-7. doi: 10.2337/diacare.18.8.1160. PMID 7587852
- [Background] Ziegler D, Hanefeld M, Ruhnau KJ, Meissner HP, Lobisch M, Schutte K, Gries FA. Treatment of symptomatic diabetic peripheral neuropathy with the anti-oxidant alpha-lipoic acid. A 3-week multicentre randomized controlled trial (ALADIN Study). Diabetologia. 1995 Dec;38(12):1425-33. doi: 10.1007/BF00400603. PMID 8786016
- [Background] Ziegler D, Hanefeld M, Ruhnau KJ, Hasche H, Lobisch M, Schutte K, Kerum G, Malessa R. Treatment of symptomatic diabetic polyneuropathy with the antioxidant alpha-lipoic acid: a 7-month multicenter randomized controlled trial (ALADIN III Study). ALADIN III Study Group. Alpha-Lipoic Acid in Diabetic Neuropathy. Diabetes Care. 1999 Aug;22(8):1296-301. doi: 10.2337/diacare.22.8.1296. PMID 10480774
- [Background] Strokov IA, Kozlova NA, Mozolevskii IuV, Miasoedov SP, Iakhno NN. [The efficacy of the intravenous administration of the trometamol salt of thioctic (alpha-lipoic) acid in diabetic neuropathy]. Zh Nevrol Psikhiatr Im S S Korsakova. 1999;99(6):18-22. Russian. PMID 10441861
- [Background] Ametov AS, Barinov A, Dyck PJ, Hermann R, Kozlova N, Litchy WJ, Low PA, Nehrdich D, Novosadova M, O'Brien PC, Reljanovic M, Samigullin R, Schuette K, Strokov I, Tritschler HJ, Wessel K, Yakhno N, Ziegler D; SYDNEY Trial Study Group. The sensory symptoms of diabetic polyneuropathy are improved with alpha-lipoic acid: the SYDNEY trial. Diabetes Care. 2003 Mar;26(3):770-6. doi: 10.2337/diacare.26.3.770. PMID 12610036
- [Background] Ruhnau KJ, Meissner HP, Finn JR, Reljanovic M, Lobisch M, Schutte K, Nehrdich D, Tritschler HJ, Mehnert H, Ziegler D. Effects of 3-week oral treatment with the antioxidant thioctic acid (alpha-lipoic acid) in symptomatic diabetic polyneuropathy. Diabet Med. 1999 Dec;16(12):1040-3. doi: 10.1046/j.1464-5491.1999.00190.x. PMID 10656234
- [Background] Dyck PJ, Kratz KM, Lehman KA, Karnes JL, Melton LJ 3rd, O'Brien PC, Litchy WJ, Windebank AJ, Smith BE, Low PA, et al. The Rochester Diabetic Neuropathy Study: design, criteria for types of neuropathy, selection bias, and reproducibility of neuropathic tests. Neurology. 1991 Jun;41(6):799-807. doi: 10.1212/wnl.41.6.799. PMID 2046920
- [Background] Dyck PJ, Karnes JL, O'Brien PC, Litchy WJ, Low PA, Melton LJ 3rd. The Rochester Diabetic Neuropathy Study: reassessment of tests and criteria for diagnosis and staged severity. Neurology. 1992 Jun;42(6):1164-70. doi: 10.1212/wnl.42.6.1164. PMID 1603343
- [Background] UK Prospective Diabetes Study Group. Tight blood pressure control and risk of macrovascular and microvascular complications in type 2 diabetes: UKPDS 38. UK Prospective Diabetes Study Group. BMJ. 1998 Sep 12;317(7160):703-13. PMID 9732337
- [Background] Reljanovic M, Reichel G, Rett K, Lobisch M, Schuette K, Moller W, Tritschler HJ, Mehnert H. Treatment of diabetic polyneuropathy with the antioxidant thioctic acid (alpha-lipoic acid): a two year multicenter randomized double-blind placebo-controlled trial (ALADIN II). Alpha Lipoic Acid in Diabetic Neuropathy. Free Radic Res. 1999 Sep;31(3):171-9. doi: 10.1080/10715769900300721. PMID 10499773
- [Derived] Ziegler D, Ametov A, Barinov A, Dyck PJ, Gurieva I, Low PA, Munzel U, Yakhno N, Raz I, Novosadova M, Maus J, Samigullin R. Oral treatment with alpha-lipoic acid improves symptomatic diabetic polyneuropathy: the SYDNEY 2 trial. Diabetes Care. 2006 Nov;29(11):2365-70. doi: 10.2337/dc06-1216. PMID 17065669